CLINICAL TRIAL: NCT05884567
Title: Effectiveness of Neck Isometric Exercises and Cervical Mobilization on Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Collaborators: Al Nafees Medical Hospital, Islamabad (Unknown); National Institute of Rehabilitation Medicine, Islamabad, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 342
Record Dates: First submitted 2023-05-13; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A single blind RCT
Who Masked: Participant
Masking Description: Just participants will have no idea in which group they are.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): neck isometric exercises will be administered at for 4 weeks and will be evaluuated at baseline, 2nd and after 4 weeks of interventions
  Interventions: Other: Isometric exercises
- control (Active Comparator): cervical mobilization will be administered at for 4 weeks and will be evaluuated at baseline, 2nd and after 4 weeks of interventions
  Interventions: Other: Mobilization

INTERVENTIONS:
Other: Isometric exercises — These exercises are used to increase muscle endurance, power and ROM
  Arms: experimental
Other: Mobilization — These exercises are used to increase ROM and used for pain reduction
  Arms: control

SUMMARY:
Effectiveness of neck isometric exercises and cervical mobilization will be compared to observe the efficacy of these techniques on cervical radiculopathy

DETAILED DESCRIPTION:
Two groups will be formed to observe the efficacy of neck isometric exercises and cervical mobilization on cervical radiculopathy by using NPRS, ROM and QoL tools.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with age between 25-50 years
* Patients referred from neuro and orthopedic departments with diagnosed cervical radiculopathy.
* Complaint of neck pain on neck bending with positive spurling's test.
* Complaint of neck pain, numbness and tingling in arm with positive spurling's test.

Exclusion Criteria:

* Cervical Trauma
* Any other orthopedic and neurological conditions of cervical spine.
* Fracture
* Malignancy

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  0 means no pain and 10 means worst pain ever
Range of motion | 4 weeks
  Goniometer will be used to assess the ranges. lower values means more limited ROM and more values means normal

CONTACTS AND LOCATIONS:
Locations (1):
- Al Nafees Medical Hospital, Islamabd, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Have not decided yet